CLINICAL TRIAL: NCT07061210
Title: An Explorative Study of HRS-2189 Combined With Adebrelimab and BP102 for Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junjie Peng, Prof., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-IIT-HRS2189-SHR1316
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-2189 + Adebrelimab + BP102 (Experimental)
  Interventions: Drug: HRS-2189; Drug: Adebrelimab; Drug: BP102

INTERVENTIONS:
Drug: HRS-2189 — HRS-2189
Drug: Adebrelimab — Adebrelimab
Drug: BP102 — BP102

SUMMARY:
To evaluate the safety and efficacy of HRS-2189 combined with Adebrelimab and BP102 in the treatment of metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1.18-75 years; 2.Histological confirmed metastatic colorectal cancer; 3.ECOG PS 0-1; 4.At least one measurable lesion (according to RECIST1.1); 5.Patients voluntarily enroll in the study.

Exclusion Criteria:

1. The patient has had other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
2. Symptomatic brain or meningeal metastases (except for those whose BMS disease is stable for at least 4 weeks);
3. Allergy to the study drug or any of its excipients;
4. Prior treatments or medications received before the first study treatment as follows:

   1. Major surgery within 28 days before treatment (tissue biopsy for diagnostic purposes is allowed).
   2. Use of immunosuppressive drugs within 7 days before treatment, excluding intranasal and inhaled corticosteroids or physiological doses of systemic steroids (i.e., no more than 10 mg/day of prednisone or an equivalent dose of other corticosteroids);
   3. Administration of immunomodulatory drugs (such as thymosin, interferon, interleukin) within 3 weeks before treatment;
   4. Vaccination with live attenuated vaccines within 28 days before treatment;
   5. Other systemic anti-tumor therapies within 28 days before treatment;
5. Any active autoimmune disease or a history of autoimmune disease with an anticipated recurrence;
6. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
7. Active infection or unexplained fever >38.5°C within 4 weeks before the first dose or on the day of the first dose (fever due to tumor may be included in the study at the investigator's discretion)；
8. Within 6 months prior to study entry, any of the following conditions: myocardial infarction, severe/unstable angina, NYHA Class 2 or higher cardiac insufficiency, or clinically significant supraventricular/ventricular arrhythmia requiring clinical intervention; poorly controlled hypertension despite medication;
9. History of severe bleeding (>30 mL per episode) within 3 months, hemoptysis (>5 mL per episode) within 1 month, or arterial/venous thrombotic events within 6 months before the first dose;
10. Inability to swallow the study drug, or presence of factors affecting drug administration and absorption such as chronic diarrhea (including but not limited to irritable bowel syndrome, Crohn's disease, ulcerative colitis) or intestinal obstruction;
11. Pregnant or breastfeeding women, or subjects of reproductive potential unwilling to use effective contraception;
12. Presence of other severe physical or laboratory abnormalities that may increase the risk of study participation, interfere with study results, or patients deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | assessed up to 1 year
  the proportion of patients with complete response or partial response, using RECIST v 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | assessed up to 1 year
  time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator
Overall survival (OS) | assessed up to 2 year
  time from enrollment to death from any cause.
Disease Control Rate (DCR) | assessed up to 1 year
  the proportion of patients with complete response, partial response or stable disease, using RECIST v 1.1.
Adverse events (AEs) | From the first drug administration to within 90 days for the last dose
  AEs are assessed by NCI-CTCAE v5.0